CLINICAL TRIAL: NCT03898284
Title: Impulse Oscillometry for Prognostication in Idiopathic Pulmonary Fibrosis
Acronym: OSCILLO
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18/OSCILLO; 2018-A02300-55 (Other: IdRCB)
Record Dates: First submitted 2019-02-26; First posted 2019-04-01 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Impulse Oscillometry; Forced Vital Capacity
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Impulse Oscillometry: Patients with Idiopathic Pulmonary Fibrosis. The objective is to determine whether another lung function technique, impulse oscillometry, is of interest to identify disease progression before changes in forced vital capacity can be ascertained.
  Interventions: Diagnostic Test: Impulse Oscillometry

INTERVENTIONS:
Diagnostic Test: Impulse Oscillometry — Impulse Oscillometry will be performed in addition to usual care

SUMMARY:
A 5-point decline of forced vital capacity expressed as % predicted, over 6 months, is the current definition of disease progression (fast decline in lung function) in idiopathic pulmonary fibrosis. There is a need for techniques allowing to characterize disease progression earlier, so that treatment may be adapted as early as possible in the lack of a response.

Hypothesis. Our hypothesis is that 3-month changes of lung function parameters measured by a novel technique, impulse oscillometry, predicts 6-month changes in forced vital capacity in idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
A 5-point decline of forced vital capacity expressed as % predicted, over 6 months, is the current definition of disease progression (fast decline in lung function) in idiopathic pulmonary fibrosis. There is a need for techniques allowing to characterize disease progression earlier, so that treatment may be adapted as early as possible in the lack of a response.

Hypothesis. Our hypothesis is that 3-month changes of lung function parameters measured by a novel technique, impulse oscillometry, predicts 6-month changes in forced vital capacity in idiopathic pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years.
* Idiopathic Pulmonary Fibrosis defined Interstitial Lung Diseases with 1) lack of any known cause for Interstitial Lung Diseases and 2) either the "definite usual interstitial pneumonia" pattern at CT scan, or the usual interstitial pneumonia (definite, probable or possible) pattern at lung biopsy, according to the Lung Function Group of the French Pulmonology Society criteria.

Exclusion Criteria:

* History of chronic obstructive airway disease.
* History of congestive heart failure.
* Emphysema-fibrosis syndrome, defined as emphysematous lesions involving >15% of the lung area at the level of the aortic arch (upper lobes).
* History of lower respiratory infection or acute respiratory failure of any cause less than 90 days before inclusion.
* Opposition to data processing.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Idiopathic Pulmonary Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Performance of the 5-Hz reactance of the respiratory system (Xsr5) variation at 3 months, for the diagnosis of rapid decline in lung function. | Baseline, 3 months, 6 months
  Receiver operating characteristics curves will be used to determine diagnostic performance.

SECONDARY OUTCOMES:
Performance of the 3-month variation in additional impulse oscillometry parameters for the diagnosis of rapid decline in lung function | Baseline, 3 months, 6 months
  Receiver operating characteristics curves will be used to determine diagnostic performance.
Performance of baseline impulse oscillometry parameters for the diagnosis of rapid decline in lung function | Baseline, 3 months, 6 months
  Receiver operating characteristics curves will be used to determine diagnostic performance.
Assess correlations between impulse oscillometry parameters and forced vital capacity | Baseline, 3 months, 6 months
  Forced vital capacity is the total amount of air exhaled during the Forced expiratory volume test (how much air a person can exhale during a forced breath)
Assess correlations between impulse oscillometry parameters and exertional dyspnea | Baseline, 3 months, 6 months
  Dyspnea is assessed by the baseline dyspnea questionnaire and the transitional dyspnea questionnaire
Assess correlations between impulse oscillometry parameters and the extent of either fibrosis or emphysema lesions on CT scans | Baseline
  Lesions are scored by trained observers.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent PLANTIER, MD-PhD, Study Director — University Hospital, Tours
Locations (4):
- France (4):
  - Respiratory Functional Explorations, University Hospital, Lille, Lille
  - Respiratory Functional Explorations, University Hospital, Nantes, Nantes
  - Department of digestive physiology, urinary, respiratory and exercise, University Hospital, Rouen, Rouen
  - Pulmonology Department, University Hospital, Tours, Tours